CLINICAL TRIAL: NCT05057897
Title: A Phase IV Open-Label, Non-Randomized, Multi-Cohort, Multicenter Study in Previously Unvaccinated Immunocompromised Adults to Determine the Immunogenicity and Safety of AZD1222 Vaccine for the Prevention of COVID-19
Brief Title: A Study of AZD1222, a Vaccine for the Prevention of COVID-19 in Immunocompromised Adults
Acronym: VICTORIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Removal of the commitment for Immune compromised study (D81111C00010) due to recruitment challenges.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D8111C00010
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19, SARS-CoV-2
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: Previously unvaccinated immunocompromised adults will be enrolled in 5 disease cohorts of approximately 60 participants each:
  1. Solid organ transplant
  2. Hematopoietic stem cell transplant
  3. Solid organ cancer patients receiving cytotoxic chemotherapy
  4. Chronic inflammatory disorders
  5. Primary immunodeficiency A sixth cohort of immunocompetent individuals will also be recruited. Participants will be allocated to the immunocompromised cohorts according to the underlying aetiology of their immunocompromised status.
  Immunocompromised participants will receive a third dose (primary vaccination series) 4 weeks or more after dose 2 with AZD1222 and will continue to be followed to the end of the study. Immunocompetent participants will be eligible to receive a third dose booster 6 months after dose 1 and will continue to be followed to the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 - immunocompromised participants with solid organ transplant (Other): Previously unvaccinated immunocompromised participants with solid organ transplant will receive a primary vaccination series with 3 IM doses of AZD1222 separated by 4 weeks and will be followed to the end of the study. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1, and the third dose will be administered 28 days after dose 2.
  Interventions: Biological: AZD1222
- Cohort 2 - immunocompromised participants with hematopoietic stem cell transplant (Other): Previously unvaccinated immunocompromised participants with hematopoietic stem cell transplant will receive a primary vaccination series with 3 IM doses of AZD1222 separated by 4 weeks and will be followed to the end of the study. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1, and the third dose will be administered 28 days after dose 2.
  Interventions: Biological: AZD1222
- Cohort 3 - immunocompromised participants with solid organ cancer receiving cytotoxic chemotherapy (Other): Previously unvaccinated immunocompromised participants with solid organ cancer receiving cytotoxic chemotherapy will receive a primary vaccination series with 3 IM doses of AZD1222 separated by 4 weeks and will be followed to the end of the study. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1, and the third dose will be administered 28 days after dose 2.
  Interventions: Biological: AZD1222
- Cohort 4 - immunocompromised participants with chronic inflammatory disorders (Other): Previously unvaccinated immunocompromised participants with chronic inflammatory disorders will receive a primary vaccination series with 3 IM doses of AZD1222 separated by 4 weeks and will be followed to the end of the study. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1, and the third dose will be administered 28 days after dose 2.
  Interventions: Biological: AZD1222
- Cohort 5 - immunocompromised participants with primary immunodeficiency (Other): Previously unvaccinated immunocompromised participants with primary immunodeficiency will receive a primary vaccination series with 3 IM doses of AZD1222 separated by 4 weeks and will be followed to the end of the study. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1, and the third dose will be administered 28 days after dose 2.
  Interventions: Biological: AZD1222
- Cohort 6 - immunocompetent participants (Other): Previously unvaccinated immunocompetent participants will receive a primary vaccination series with 2 IM doses of AZD1222 separated by 4 weeks, followed by a booster dose of AZD1222 administered 6 months after the first dose. The first dose will be administered on Day 1, the second dose will be administered 28 days after dose 1. Participants will receive a third dose booster 6 months after dose 1 and will continue to be followed to the end of the study.
  Interventions: Biological: AZD1222

INTERVENTIONS:
Biological: AZD1222 — 10 mM histidine, 7.5% (w/v) sucrose, 35 mM sodium chloride, 1 mM magnesium chloride, 0.1% (w/v) polysorbate 80, 0.1 mM edetate disodium, 0.5% (w/v) ethanol, at pH 6.6

SUMMARY:
The aim of this study is to assess the immunogenicity and safety of AZD1222 for prevention of COVID-19 in immunocompromised adults.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the immunogenicity and safety of AZD1222, AstraZeneca's approved ChAdOx1 vector vaccine against SARS-CoV-2, in SARS-CoV-2 seronegative immunocompromised individuals who are unvaccinated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ≥ 18 years at the time of signing the informed consent.
2. Cohort specific inclusion criteria:

Solid organ transplant

* Participants with heart, lung, kidney, or liver transplant, and are stable on immunosuppressants (defined as no change in dose in the previous 4 weeks).

Hematopoietic stem cell transplant

* Participants with autologous (up to 6 months after transplantation) or allogeneic stem cell transplant who are immunosuppressed, with no evidence of active graft-versushost disease, at least one month after the procedure.

Cancer patients on chemotherapy

* Participants with solid tumors (except breast cancer), histologically diagnosed, who were undergoing intravenous cytotoxic chemotherapy within the last 6 months, who received at least 1 cycle prior to cytotoxic chemotherapy, and have a life expectancy of longer than 3 months.

Chronic inflammatory conditions

* Participants with chronic inflammatory conditions, including those on immunosuppressant medications, can be recruited. The following conditions are specifically excluded: multiple sclerosis and peripheral demyelinating disease.

Primary immune deficiency

* Examples include combined granulomatous disorder, SCID, common variable immunodeficiency.

Immunocompetent:

* No confirmed or suspected immunosuppressive or immunodeficient state.
* No use of immunosuppressant medication within the past 1 month (≥ 20 mg per day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days within 30 days prior to administration of AZD1222). The following exceptions are permitted: topical/inhaled steroids or short-term oral steroids (course lasting ≤ 14 days).
* No receipt of immunoglobulins and/or any blood products within 3 months prior to administration of AZD1222 or expected receipt during the period of study follow up.
* No severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness, as judged by the Investigator.

Exclusion Criteria:

1. History of allergic disease or reactions likely to be exacerbated by any component of AZD1222.
2. Active infection with SARS-CoV-2 as confirmed locally by nucleic acid amplification test (e.g. RT-PCR).
3. Known current or past laboratory-confirmed SARS-CoV-2 infection.
4. Significant infection or other acute illness, including fever (temperature > 37.8°C) on the day prior to or day of first dosing.
5. Thrombocytopenia with platelet count ≤ 75,000 x 109/microliter based on complete blood count test at screening visit.
6. HIV-positive participants based on a positive ELISA test performed at screening visit.
7. History of cerebral venous sinus thrombosis (CVST).
8. Receipt of any vaccine (licensed or investigational) within 30 days prior to and after administration of AZD1222.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Muang
- Research Site, Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111C00010&attachmentIdentifier=41c47426-8c12-43ce-a602-6e2f7a216256&fileName=D8111C00010-CSR_synopsis_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase IV open-label study was conducted in previously unvaccinated immunocompromised adult participants at 4 sites in Ukraine and Thailand between 31 Jan 2022 and 19 Apr 2023. The study was terminated prematurely due to recruitment challenges, resulting in low sample sizes, especially in the immunocompromised cohorts. Hence, analyses were streamlined.
Pre-assignment Details: This study consisted of a screening period (up to 7 days) and a vaccination/follow-up period (up to 365 days). The study was planned to involve a total of 6 cohorts: 5 immunocompromised cohorts (including participants with solid organ transplant, hematopoietic stem cell transplant, solid organ cancer participants receiving cytotoxic chemotherapy, chronic inflammatory disorders and primary immunodeficiency) and 1 immunocompetent cohort.
Groups:
- Immunocompromised Cohort: Participants received 3 IM doses of AZD1222 5 × 10^10 vp on Days 1, 29 and 57.
- Immunocompetent Cohort: Participants received 3 IM doses of AZD1222 5 × 10^10 vp on Days 1, 29 and 183.
Period: Overall Study
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Started | 11 | 23
Received 1 Dose | 11 | 23
Received 2 Doses | 9 | 20
Received 3 Doses | 6 | 13
Completed | 8 | 21
Not Completed | 3 | 2
Not completed — Site closure | 2 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis set consisted of all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort | Total
Number analyzed (Participants) | 11 | 23 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 21 | 28
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 4 | 12 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 4
  Asian | 9 | 21 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 11 | 23 | 34

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibodies (nAb) Post 2-Dose Primary Vaccination of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The GMT was calculated as the antilogarithm of Σ (base 2 log transformed titer/n), that is (i.e.), as the antilogarithm transformation of the mean of the log-transformed titer, where n is the number of participants with titer information.
Time Frame: Days 29 and 57
Population: The Immunogenicity Analysis set (IAS) consisted of all participants in the Safety Analysis set who had at least 1 baseline and post-baseline record in immunogenicity data and no protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response. Only those participants with data available were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 9 | 18
1/dilution
  Day 29 | 47.7 [14.9 to 152.6] | 67.9 [31.5 to 146.3]
  Day 57: number analyzed (Participants) | 8 | 14
  Day 57 | 122.0 [31.0 to 479.7] | 166.5 [96.2 to 288.1]

2. Primary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 nAb Post 2-Dose Primary Vaccination of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post doses 1 and 2) to SARS-CoV-2 nAb of AZD1222 as measured by pseudo-neutralization assay is reported. The 2-sided 95% CI was calculated using Clopper-Pearson methodology.
Time Frame: Days 29 and 57
Population: The IAS consisted of all participants in the Safety Analysis set who had at least 1 baseline and post-baseline record in immunogenicity data and no protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response. Only those participants with data available were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 9 | 18
percentage of participants
  Day 29 | 22.2 [2.80 to 60.00] | 44.4 [21.50 to 69.20]
  Day 57: number analyzed (Participants) | 8 | 14
  Day 57 | 62.5 [24.50 to 91.50] | 92.9 [66.10 to 99.80]

3. Primary Outcome: GMT for SARS-CoV-2 Anti-Spike Binding Antibodies Post 2-Dose Primary Vaccination of AZD1222 as Measured by Meso Scale Discovery (MSD) Serology Assay
Description: The GMT was calculated as the antilogarithm of Σ (base 2 log transformed titer/n), i.e, as the antilogarithm transformation of the mean of the log-transformed titer, where n is the number of participants with titer information.
Time Frame: Days 29 and 57
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units (AU)/milliliter (mL)
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 9 | 18
arbitrary units (AU)/milliliter (mL)
  Day 29 | 3997.2 [1285.9 to 12425.7] | 19134.7 [10824.2 to 33825.8]
  Day 57: number analyzed (Participants) | 8 | 14
  Day 57 | 13262.8 [1617.8 to 108732.5] | 28320.9 [20744.6 to 38664.1]

4. Primary Outcome: Percentage of Participants With Seroresponse to Anti-Spike Binding Antibodies of a 2-Dose Primary Vaccination of AZD1222 as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post doses 1 and 2) to anti-spike binding antibodies of AZD1222 as measured by MSD serology assay is reported. The 2-sided 95% CI was calculated using Clopper-Pearson methodology.
Time Frame: Days 29 and 57
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 9 | 18
percentage of participants
  Day 29 | 88.9 [51.80 to 99.70] | 100 [81.50 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100.
  Day 57: number analyzed (Participants) | 8 | 14
  Day 57 | 75.0 [34.90 to 96.80] | 100 [76.80 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100.

5. Secondary Outcome: GMT for SARS-CoV-2 nAb Post Second Dose of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The GMT was calculated as the antilogarithm of Σ (base 2 log transformed titer/n), i.e., as the antilogarithm transformation of the mean of the log-transformed titer, where n is the number of participants with titer information. The ratio of SARS-CoV-2 specific GMT titers 28 days post Dose 2 of AZD1222 was calculated as the ratio of the titer levels in the immunocompromised cohort to the immunocompetent cohort.
Time Frame: Day 57
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 8 | 14
1/dilution | 122.0 [31.0 to 479.7] | 166.5 [96.2 to 288.1]
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 57 (28 days post Dose 2); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; GMT Ratio = 0.73, 95% CI 2-sided [0.18 to 3.01] — The GMT ratio was calculated as the ratio of the titer levels in the immunocompromised cohort to the immunocompetent cohort

6. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 nAb Post Second Dose of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post Dose 2) to SARS-CoV-2 nAb of AZD1222 as measured by pseudo-neutralization assay is reported, and the 2-sided 95% CI was calculated using Clopper-Pearson methodology. The difference in seroresponse 28 days post Dose 2 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort), and the 2-sided 95% CI was calculated using the Newcombe score without continuity correction.
Time Frame: Day 57
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 8 | 14
percentage of participants | 62.5 [24.50 to 91.50] | 92.9 [66.10 to 99.80]
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 57 (28 days post Dose 2); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; The 2-sided 95% CI was calculated using the Newcombe score without continuity correction; Difference in Seroresponse = -30.36, 95% CI 2-sided [-62.82 to 3.69] — The difference in seroresponse 28 days post Dose 2 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort)

7. Secondary Outcome: GMT for SARS-CoV-2 Anti-Spike Binding Antibodies Post Second Dose of AZD1222 as Measured by MSD Serology Assay
Description: as for outcome 5
Time Frame: Day 57
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units (AU)/milliliters (mL)
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 8 | 14
arbitrary units (AU)/milliliters (mL) | 13262.8 [1617.8 to 108732.5] | 28320.9 [20744.6 to 38664.1]
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 57 (28 days post Dose 2); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; GMT Ratio = 0.47, 95% CI 2-sided [0.06 to 3.86] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Anti-Spike Binding Antibodies Post Second Dose of AZD1222 as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post Dose 2) to SARS-CoV-2 nAb of AZD1222 as measured by MSD Serology assay is reported, and the 2-sided 95% CI was calculated using Clopper-Pearson methodology. The difference in seroresponse 28 days post Dose 2 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort), and the 2-sided 95% CI was calculated using the Newcombe score without continuity correction.
Time Frame: Day 57
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 8 | 14
percentage of participants | 75.0 [34.90 to 96.80] | 100 [76.80 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100.
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 57 (28 days post Dose 2); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; The 2-sided 95% CI was calculated using the Newcombe score without continuity correction; Difference in Seroresponse = -25.00, 95% CI 2-sided [-59.07 to 2.97] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: GMT for SARS-CoV-2 nAb Post Third Dose of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The GMT was calculated as the antilogarithm of Σ (base 2 log transformed titer/n), i.e., as the antilogarithm transformation of the mean of the log-transformed titer, where n is the number of participants with titer information. The ratio of SARS-CoV-2 specific GMT titers 28 days post Dose 3 of AZD1222 was calculated as the ratio of the titer levels in the immunocompromised cohort to the immunocompetent cohort.
Time Frame: Day 85 for immunocompromised cohort and Day 211 for immunocompetent cohort
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 2 | 12
1/dilution | 224.5 [13.6 to 3717.8] | 710.3 [345.3 to 1461.3]
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 85 Immunocompromised / Day 211 Immunocompetent (28 days post Dose 3); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; GMT Ratio = 0.32, 95% CI 2-sided [0.12 to 0.80] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 nAb Post Third Dose of AZD1222 as Measured by Pseudo-neutralization Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post dose 3) to SARS-CoV-2 nAb of AZD1222 as measured by pseudo-neutralization assay is reported, and the 2-sided 95% CI was calculated using Clopper-Pearson methodology. The difference in seroresponse 28 days post Dose 3 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort).
Time Frame: Day 85 for immunocompromised cohort and Day 211 for immunocompetent cohort
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 2 | 12
percentage of participants | 100 [15.80 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100. | 100 [73.50 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100.
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 85 Immunocompromised / Day 211 Immunocompetent (28 days post Dose 3); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; Due to everyone in both cohorts being a seroresponder, the confidence interval (CI) around the difference is not estimable; Difference in Seroresponse = 0 — The difference in seroresponse 28 days post Dose 3 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort)

11. Secondary Outcome: GMT for SARS-CoV-2 Anti-Spike Binding Antibodies Post Third Dose of AZD1222 as Measured by MSD Serology Assay
Description: as for outcome 9
Time Frame: Day 85 for immunocompromised cohort and Day 211 for immunocompetent cohort
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units (AU)/milliliters (mL)
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 2 | 12
arbitrary units (AU)/milliliters (mL) | 48303.4 [4118.7 to 566496.7] | 86462.9 [47538.3 to 157259.2]
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 85 Immunocompromised / Day 211 Immunocompetent (28 days post Dose 3); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; GMT Ratio = 0.56, 95% CI 2-sided [0.25 to 1.25] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Percentage of Participants With Seroresponse to Anti-Spike Binding Antibodies Post Third Dose of AZD1222 as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. The percentage of participants with a post-intervention seroresponse (>=4-fold rise in titers from baseline value to 28 days post dose 3) to anti-spike binding antibodies of AZD1222 as measured by MSD serology assay is reported, and the 2-sided 95% CI was calculated using Clopper-Pearson methodology. The difference in seroresponse 28 days post Dose 3 of AZD1222 was calculated as (seroresponse rate of immunocompromised cohort) - (seroresponse rate of immunocompetent cohort).
Time Frame: Day 85 for immunocompromised cohort and Day 211 for immunocompetent cohort
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
Number analyzed (Participants) | 2 | 12
percentage of participants | 100 [15.80 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100. | 100 [73.50 to NA] — Due to the point estimate of 100% being on the boundary (0% or 100%), only the lower bound of the confidence interval (CI) is meaningful. To reflect this, the upper bound is reported as NA instead of 100.
Statistical Analysis 1: Comparison: Immunocompromised Cohort vs Immunocompetent Cohort; Day 85 Immunocompromised / Day 211 Immunocompetent (28 days post Dose 3); Test type: Other — Descriptive only. Analysis conducted at request of clinicaltrials.gov; [statistical method as in outcome 10, analysis 1]; Difference in Seroresponse = 0 — [estimate comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from start of treatment administration (Day 1) up to end of study (approximately 15 months)
Description: The Safety Analysis set consisted of all participants who received at least 1 dose of study treatment.
Arm/Group | Immunocompromised Cohort | Immunocompetent Cohort
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/11 | 4/23
Other Adverse Events (participants affected / at risk) | 7/11 | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunocompromised Cohort (N=11) | Immunocompetent Cohort (N=23)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunocompromised Cohort (N=11) | Immunocompetent Cohort (N=23)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to recruitment challenges, resulting in low sample sizes, especially in the immunocompromised cohorts. Hence, all outcome measures, including comparisons between cohorts, should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT05057897/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT05057897/SAP_001.pdf